CLINICAL TRIAL: NCT01155466
Title: A Phase 3, 12-Week, Double-Blind, Double-Dummy, Placebo- and Active-Controlled Efficacy and Safety Study of Preladenant in Subjects With Moderate to Severe Parkinson's Disease (Phase 3;Protocol No. P04938)
Brief Title: A Placebo- and Active Controlled Study of Preladenant in Subjects With Moderate to Severe Parkinson's Disease (P04938)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P04938; 2009-015161-31 (EudraCT Number); CTRI/2011/07/001896 (Registry Identifier: CTRI); MK-3814-015 (Other: Merck Protocol Number)
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Parkinson Disease
Keywords: Idiopathic Parkinson Disease; Idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — 2-(2-furanyl)-7-(2-(4-(4-(2-methoxyethoxy)phenyl)-1-piperazinyl)ethyl)-7H-pyrazolo(4,3-e)(1,2,4)triazolo(1,5-c)pyrimidine-5-amine; Tablets; rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Preladenant 2 mg (Experimental): Preladenant 2 mg tablet + placebo to rasagiline capsule in AM and preladenant 2 mg tablet in PM for 12 weeks
  Interventions: Drug: Preladenant 2 mg tablet; Drug: Placebo to Rasagiline capsule
- Preladenant 5 mg (Experimental): Preladenant 5 mg tablet + placebo to rasagiline capsule in AM and preladenant 5 mg tablet in PM for 12 weeks
  Interventions: Drug: Preladenant 5 mg tablet; Drug: Placebo to Rasagiline capsule
- Preladenant 10 mg (Experimental): Preladenant 10 mg tablet + placebo to rasagiline capsule in AM and preladenant 10 mg tablet in PM for 12 weeks
  Interventions: Drug: Preladenant 10 mg tablet; Drug: Placebo to Rasagiline capsule
- Placebo (Placebo Comparator): Placebo to preladenant tablet + placebo to rasagiline capsule in AM and placebo to preladenant tablet in PM for 12 weeks
  Interventions: Drug: Placebo to Preladenant Tablet; Drug: Placebo to Rasagiline capsule
- Rasagiline 1 mg (Active Comparator): Rasagiline 1 mg capsule + placebo to preladenant tablet in AM and placebo to preladenant tablet in PM for 12 weeks
  Interventions: Drug: Placebo to Preladenant Tablet; Drug: Rasagiline 1 mg capsule

INTERVENTIONS:
Drug: Preladenant 2 mg tablet — one 2 mg tablet orally twice daily
  Other Names: SCH 420814
  Arms: Preladenant 2 mg
Drug: Preladenant 5 mg tablet — one 5 mg tablet orally twice daily
  Other Names: SCH 420814
  Arms: Preladenant 5 mg
Drug: Preladenant 10 mg tablet — one 10 mg tablet orally twice daily
  Other Names: SCH 420814
  Arms: Preladenant 10 mg
Drug: Placebo to Preladenant Tablet — one tablet orally twice daily
  Arms: Placebo; Rasagiline 1 mg
Drug: Rasagiline 1 mg capsule — one 1 mg capsule orally in AM
  Other Names: Azilect
  Arms: Rasagiline 1 mg
Drug: Placebo to Rasagiline capsule — one capsule orally in AM
  Arms: Placebo; Preladenant 10 mg; Preladenant 2 mg; Preladenant 5 mg

SUMMARY:
When a patient with Parkinson's disease (PD) is initially treated with L-dopa or dopamine agonists, the symptoms of PD improve or disappear. After several years of taking L dopa or dopamine agonists, patients notice that their PD medications wear off sooner than when they first started taking them. This "wearing off" is characterized by the return of symptoms (i.e., tremor, slowness, and rigidity) and may occur over the course of a few minutes to an hour. When a patient's PD symptoms have returned, the patient is said to be in the "off" state. When the patient takes another dose of medication, and his/her PD symptoms improve or resolve, the patient is said to be in the "on" state. Antagonism of adenosine Type 2a receptors (A2a) may provide relief of PD symptoms. This trial will test the hypothesis that A2a receptor antagonism can lead to improvement in the function of PD participants taking a stable dose of L-dopa, as measured by a reduction in "off" time.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of moderate to severe idiopathic Parkinson's disease.
* Must have received prior therapy with L dopa for approximately 1 or more years immediately before Screening and must continue to have a beneficial clinical response to L dopa
* Must have been on a stable dopaminergic treatment regimen for at least the 5 weeks immediately before Randomization. Participants receiving other adjunctive treatments (eg, dopamine agonists, anticholinergics, entacapone) or taking only L dopa are permitted, provided the treatment regimen has been taken for at least 5 weeks prior to randomization
* Must be experiencing motor fluctuations with or without dyskinesias within the 4 weeks immediately before Screening, must be experiencing a minimum of 2 hours/day of "off" time, and have a Hoehn & Yahr stage between 2.5 and 4 when in the "on" state
* Must be capable of maintaining an accurate and complete symptom diary and to adhere to dose and visit schedules with or without the help of a caregiver
* Must have results of a physical examination and screening clinical laboratory tests clinically acceptable to the investigator
* If sexually active or plan to be sexually active agree to use a highly effective method of birth control while in the study and for 2 weeks after the last dose of study drug. Males must also not donate sperm during the trial within 2 weeks after the last dose of study drug

Exclusion Criteria:

* Must not have a form of drug induced or atypical parkinsonism, a cognitive impairment, bipolar disorder, untreated major depressive disorder, schizophrenia, or other psychotic disorder; history of exposure to a known neurotoxin, or any neurological features not consistent with the diagnosis of PD as assessed by the investigator
* Must not have a history of repeated strokes or head injuries, or a stroke within 6 months of Screening
* Must not have poorly-controlled diabetes or abnormal renal function
* Must not have had surgery for their PD
* Must not be at imminent risk of self-harm or harm to others
* Must not have sleep attacks or compulsive behavior that would interfere with the integrity of the trial or would pose a risk to the subject in participating in the trial
* Must not have a systolic blood pressure (BP) ≥150 mm Hg OR diastolic BP ≥95 mm Hg at Screening
* Must not have had any clinically significant cardiovascular event or procedure for 6 months prior to study start, including, but not limited to, myocardial infarction, angioplasty, unstable angina, or heart failure; and must not have heart failure staged New York Heart Association Class III or IV
* Must not have an alanine aminotransferase (ALT) or aspartate amino transferase (AST) ≥3 x the upper limit of normal (ULN) or total bilirubin (T-BIL) ≥1.5 x ULN
* Must not have a history of serologically confirmed hepatic dysfunction (defined as viral infection [Hepatitis B or C; Epstein Barr virus (EBV); cytomegalovirus (CMV)]) or a history of diagnosis of drug or alcohol induced hepatic toxicity or frank hepatitis
* Must not have a history within the past 5 years of a primary or recurrent malignant disease with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or in situ prostate cancer with a normal prostate-specific antigen (PSA) post resection
* Must not have received certain prespecified medications or ingested high tyramine-containing aged cheeses (eg, Stilton) for a prespecified time window before the trial, during the trial, and for 2 weeks after the trial
* Must not have an average daily consumption of more than three 4 ounce glasses (118 mL) of wine or the equivalent
* Must not have a severe or ongoing unstable medical condition (eg, any form of clinically significant cardiac disease, symptomatic orthostatic hypotension, seizures, or alcohol/drug dependence)
* Must not have allergy/sensitivity to investigational product(s) or its/their excipients
* A female subject must not be breast-feeding, considering breast-feeding, pregnant, or intending to become pregnant
* Must not have used preladenant ever, or any investigational drugs within 90 days immediately before Screening

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 778 (Actual)
Dates: Start 2010-07-14 (Actual); Primary Completion 2012-12-20 (Actual); Study Completion 2012-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Hauser RA, Stocchi F, Rascol O, Huyck SB, Capece R, Ho TW, Sklar P, Lines C, Michelson D, Hewitt D. Preladenant as an Adjunctive Therapy With Levodopa in Parkinson Disease: Two Randomized Clinical Trials and Lessons Learned. JAMA Neurol. 2015 Dec;72(12):1491-500. doi: 10.1001/jamaneurol.2015.2268. PMID 26523919
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P04938&kw=P04938&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total 1076 participants were screened and 778 were randomized.
Period: Overall Study
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo | Rasagiline 1 mg
Started | 156 | 155 | 156 | 155 | 156
Treated | 154 | 153 | 153 | 155 | 154
Completed | 134 (Completed treatment phase) | 130 (Completed treatment phase) | 136 (Completed treatment phase) | 134 (Completed treatment phase) | 129 (Completed treatment phase)
Not Completed | 22 | 25 | 20 | 21 | 27
Not completed — Adverse Event | 13 | 15 | 6 | 17 | 18
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 7 | 5 | 9 | 4 | 4
Not completed — Protocol Violation | 0 | 0 | 2 | 0 | 1
Not completed — Administrative | 0 | 3 | 0 | 0 | 0
Not completed — Randomized not treated | 2 | 2 | 3 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo | Rasagiline 1 mg | Total
Number analyzed (Participants) | 156 | 155 | 156 | 155 | 156 | 778
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (9.2) | 62.6 (8.5) | 63.6 (8.4) | 63.0 (8.4) | 63.8 (9.0) | 62.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 76 | 61 | 77 | 61 | 332
  Male | 99 | 79 | 95 | 78 | 95 | 446

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean "Off" Time
Description: The "on" state is defined as the period of time during which a patient's symptoms of PD improve or disappear following treatment with L-dopa or dopamine agonists. The "off" state is defined as the period of time characterized by the return of symptoms (i..e. tremor, slowness, and rigidity) following treatment with L-dopa or dopamine agonists. Study participants reported their symptoms at half-hour intervals as "off", "on", or "asleep" on their daily diary for 3 days before randomization (baseline) and for the 3 days immediately before their Week-12 visit. The mean change from baseline in "off" time was based on a constrained longitudinal data analysis with treatment, time, and treatment-by-time interaction as fixed effects and subject as random effect.
Time Frame: Baseline and Week 12
Population: The number of randomized and treated participants with at least one post baseline value.
Measure: Mean (Standard Error); unit: Hours/day
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo | Rasagiline 1 mg
Number analyzed (Participants) | 152 | 149 | 149 | 151 | 152
Hours/day | -0.9 (0.21) | -0.9 (0.21) | -0.8 (0.21) | -0.8 (0.21) | -1.1 (0.21)
Statistical Analysis 1: Comparison: Preladenant 10 mg vs Placebo; Test type: Superiority or Other; p = 0.8700, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.62 to 0.53] — The estimated parameter is the difference in the estimated mean change from baseline in mean "off" time for preladenant 10 mg - placebo

2. Primary Outcome: Numberof Participants With Systolic Blood Pressure >=180 mm Hg
Description: The number of participants with Systolic Blood Pressure >=180 mm Hg was reported.
Time Frame: Up to Week 14
Population: The number of participants who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo | Rasagiline 1 mg
Number analyzed (Participants) | 154 | 153 | 153 | 155 | 154
Participants | 1 (0.21) | 1 (0.21) | 3 (0.21) | 1 (0.21) | 0 (0.21)

3. Primary Outcome: Number of Participants With Diastolic Blood Pressure >=105 mm Hg
Description: The number of participants with Diastolic Blood Pressure >=105 mm Hg was reported.
Time Frame: Up to Week 14
Population: The number of participants who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo | Rasagiline 1 mg
Number analyzed (Participants) | 154 | 153 | 153 | 155 | 154
Participants | 3 (0.21) | 4 (0.21) | 9 (0.21) | 7 (0.21) | 4 (0.21)
Statistical Analysis 1: Comparison: Preladenant 2 mg vs Placebo; Test type: Superiority or Other; p = 0.899, Miettinen & Nurminen; Risk Difference (RD) = -2.6, 95% CI 2-sided [-7.3 to 1.6] — The estimated parameter is the difference in the percentage of participants with diastolic blood pressure >=105 mm Hg for preladenant 2 mg - placebo
Statistical Analysis 2: Comparison: Preladenant 5 mg vs Placebo; Test type: Superiority or Other; p = 0.815, Miettinen & Nurminen; Risk Difference (RD) = -1.9, 95% CI 2-sided [-6.8 to 2.6] — The estimated parameter is the difference in the percentage of participants with diastolic blood pressure >=105 mm Hg for preladenant 5 mg - placebo
Statistical Analysis 3: Comparison: Preladenant 10 mg vs Placebo; Test type: Superiority or Other; p = 0.295, Miettinen & Nurminen; Risk Difference (RD) = 1.4, 95% CI 2-sided [-3.9 to 6.9] — The estimated parameter is the difference in the percentage of participants with diastolic blood pressure >=105 mm Hg for preladenant 10 mg - placebo

4. Primary Outcome: Number of Participants With Alanine Aminotransferase >=3 Times the Upper Limit of Normal
Description: The number of participants with alanine aminotransferase >=3 times the upper limit of normal and a >=10% increase was reported.
Time Frame: Up to Week 14
Population: The number of participants who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo | Rasagiline 1 mg
Number analyzed (Participants) | 154 | 153 | 153 | 155 | 154
Participants | 1 (0.21) | 1 (0.21) | 1 (0.21) | 1 (0.21) | 0 (0.21)

5. Primary Outcome: Number of Participants With Aspartate Aminotransferase >=3 Times the Upper Limit of Normal
Description: The number of participants with aspartate aminotransferase >=3 times the upper limit of normal and a >=10% increase was reported.
Time Frame: Up to Week 14
Population: The number of participants who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo | Rasagiline 1 mg
Number analyzed (Participants) | 154 | 153 | 153 | 155 | 154
Participants | 1 (0.21) | 1 (0.21) | 1 (0.21) | 0 (0.21) | 0 (0.21)

6. Primary Outcome: Percentage of Participants With Suicidality
Description: The percentage of participants with suicidality using the Columbia - Suicide Severity Rating Scale (C-SSRS) was reported. The C-SSR was used in this study only for the purpose of safety monitoring by measuring the incidence of different types of suicidality categories during treatment. The assessment was done by the nature of the responses, not by a numbered scale. Participants who reported at least one occurrence of suicidal behavior or suicidal ideation were counted as having experienced suicidality. Suicidal behavior included suicide attempt, aborted attempt, interrupted attempt, or preparatory behavior. Suicidal ideation included a wish to die or active suicidal thought with or without method, intent or plan.
Time Frame: Up to Week 12
Population: The number of participants who received at least one dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo | Rasagiline 1 mg
Number analyzed (Participants) | 154 | 153 | 153 | 155 | 154
Percentage of participants | 2.6 (0.21) | 2.6 (0.21) | 0.7 (0.21) | 3.2 (0.21) | 0.6 (0.21)
Statistical Analysis 1: Comparison: Preladenant 2 mg vs Placebo; Test type: Superiority or Other; p = 0.629, Miettinen & Nurminen; Risk Difference (RD) = -0.6, 95% CI 2-sided [-5.1 to 3.7] — The estimated parameter is the difference in the percentage of participants with suicidality for preladenant 2 mg - placebo
Statistical Analysis 2: Comparison: Preladenant 5 mg vs Placebo; Test type: Superiority or Other; p = 0.625, Miettinen & Nurminen; Risk Difference (RD) = -0.6, 95% CI 2-sided [-5.1 to 3.7] — The estimated parameter is the difference in the percentage of participants with suicidality for preladenant 5 mg - placebo
Statistical Analysis 3: Comparison: Preladenant 10 mg vs Placebo; Test type: Superiority or Other; p = 0.948, Miettinen & Nurminen; Risk Difference (RD) = -2.6, 95% CI 2-sided [-6.8 to 0.7] — The estimated parameter is the difference in the percentage of participants with suicidality for preladenant 10 mg - placebo

7. Primary Outcome: Change From Baseline at Week 12 in Epworth Sleepiness Scale (ESS)
Description: The ESS is a self-administered questionnaire providing a measure of a person's general level of daytime sleepiness, or their average sleep propensity in daily life. The scale consists of 8 situations in which the participant rates their tendency to become sleepy on a scale of 0=no chance of dozing to 3=high chance of dozing. The overall score is the sum of the scores for the 8 situations for a minimum of 0 and a maximum of 24.
Time Frame: Baseline and Week 12
Population: The number of participants who received at least one dose of study drug and had baseline and Week 12 data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo | Rasagiline 1 mg
Number analyzed (Participants) | 127 | 121 | 132 | 127 | 121
Scores on a scale | -0.3 (3.4) | -0.1 (3.1) | 0.0 (3.5) | -0.3 (3.1) | 0.1 (3.5)
Statistical Analysis 1: Comparison: Preladenant 2 mg vs Placebo; Test type: Superiority or Other; p = 0.7044, Constrained longitudinal data analysis; Risk Difference (RD) = 0.1, 95% CI 2-sided [-0.61 to 0.90] — The estimated parameter is the difference in the change from baseline in mean ESS score for preladenant 2 mg - placebo
Statistical Analysis 2: Comparison: Preladenant 5 mg vs Placebo; Test type: Superiority or Other; p = 0.3439, Constrained longitudinal data analysis; Risk Difference (RD) = 0.4, 95% CI 2-sided [-0.4 to 1.14] — The estimated parameter is the difference in the change from baseline in mean ESS score for preladenant 5 mg - placebo
Statistical Analysis 3: Comparison: Preladenant 10 mg vs Placebo; Test type: Superiority or Other; p = 0.3941, Constrained longitudinal data analysis; Risk Difference (RD) = 0.3, 95% CI 2-sided [-0.43 to 1.08] — The estimated parameter is the difference in the change from baseline in mean ESS score for preladenant 10 mg - placebo

8. Secondary Outcome: Percentage of Participants With >30% Change (Reduction) From Baseline at Week 12 in Mean "Off" Time
Description: The "on" state is defined as the period of time during which a patient's symptoms of PD improve or disappear following treatment with L-dopa or dopamine agonists. The "off" state is defined as the period of time characterized by the return of symptoms (i..e. tremor, slowness, and rigidity) following treatment with L-dopa or dopamine agonists. Study participants reported their symptoms at half-hour intervals as "off", "on", or "asleep" on their daily diary for 3 days before randomization and for the 3 days immediately before their Week-12 visit.
Time Frame: Baseline and Week 12
Population: The number of randomized and treated participants with a Week 12 value.
Measure: Number; unit: Percentage of participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo | Rasagiline 1 mg
Number analyzed (Participants) | 125 | 122 | 131 | 131 | 121
Percentage of participants | 30.4 | 33.6 | 35.1 | 32.8 | 33.9
Statistical Analysis 1: Comparison: Preladenant 10 mg vs Placebo; Test type: Superiority or Other; p = 0.983, Mixed Models Analysis; Odds ratio was calculated for all randomized and treated participants with at least 1 post treatment value; Odds Ratio (OR) = 0.994, 95% CI 2-sided [0.597 to 1.657] — Confidence intervals and P-values were based on a generalized linear mixed model with baseline average "off" time as a covariate and treatment-by-time interaction as fixed effect and participant as random effect

9. Secondary Outcome: Change From Baseline at Week 12 in Mean "On" Time Without Troublesome Dyskinesia
Description: When a participant is "on" without dyskinesias, parkinsonian symptoms have dissipated and the participant is experiencing no uncontrollable extraneous movements. Study participants reported their parkinsonian symptoms at half-hour intervals as "off", "on without dyskinesia", "on with non-troublesome dyskinesia", "on with troublesome dyskinesia", or "asleep" on their daily diary for 3 days before randomization and for the 3 days immediately before their Week-12 visit. The mean change from baseline in "on without troublesome dyskinesia" time was based on a constrained longitudinal data analysis with treatment, time, and treatment-by-time interaction as fixed effects and subject as random effect.
Time Frame: Baseline and Week 12
Population: The number of randomized and treated participants with at least one post baseline value.
Measure: Mean (Standard Error); unit: Hours/day
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo | Rasagiline 1 mg
Number analyzed (Participants) | 152 | 149 | 149 | 151 | 152
Hours/day | 0.8 (0.24) | 0.9 (0.24) | 0.5 (0.23) | 0.4 (0.24) | 0.7 (0.24)
Statistical Analysis 1: Comparison: Preladenant 10 mg vs Placebo; Test type: Superiority or Other; p = 0.6405, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.49 to 0.80] — The estimated parameter is the difference in the estimated change from baseline in "on" time without troublesome dyskinesias for preladenant 10 mg - placebo

ADVERSE EVENTS:
Time Frame: All adverse events: up to Week 14; serious adverse events: up to 30 days after the last dose of study drug (up to Week 16)
Description: The safety population included all participants who received at least one dose of study drug
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo | Rasagiline 1 mg
Serious Adverse Events (participants affected / at risk) | 5/154 | 4/153 | 5/153 | 6/155 | 9/154
Other Adverse Events (participants affected / at risk) | 18/154 | 20/153 | 29/153 | 34/155 | 25/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 2 mg (N=154) | Preladenant 5 mg (N=153) | Preladenant 10 mg (N=153) | Placebo (N=155) | Rasagiline 1 mg (N=154)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periproctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia malignant (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 2 mg (N=154) | Preladenant 5 mg (N=153) | Preladenant 10 mg (N=153) | Placebo (N=155) | Rasagiline 1 mg (N=154)
Constipation (Gastrointestinal disorders) | 5 (5) | 5 (5) | 16 (17) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 2 (2) | 8 (8) | 1 (1)
Dyskinesia (Nervous system disorders) | 5 (5) | 10 (13) | 7 (7) | 8 (9) | 21 (23)
Headache (Nervous system disorders) | 7 (7) | 3 (4) | 7 (7) | 16 (17) | 4 (4)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 8 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation with regard to proprietary information, accuracy, fair balance, and compliance.